CLINICAL TRIAL: NCT02177383
Title: Scientific Basis of the Action of Foods Rich in Essential Fatty Acids on the Expression of Antioxidant Genes and Athletic Performance
Brief Title: Action of Essential Fatty Acids on the Expression of Antioxidant Genes and Athletic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Antoni Pons, Professor, University of the Balearic Islands
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IB 994/08 PI
Record Dates: First submitted 2014-06-17; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Oxidative Stress; Exercise; Training Season; Antioxidant Capabilities; Athletic Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Docosahexaenoic acid (Experimental): 1 liter/day of one experimental beverage (containing 0.2% olive oil + 0.6% DHA-S Martek) provides 1.14 g DHA/daily
  Interventions: Dietary Supplement: Docosahexaenoic acid diet supplementation
- Olive oil (Placebo Comparator): 1 liter/day of placebo beverage (containing 0.8% olive oil)
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid diet supplementation — Nine soccer players (19 and 22 years old) took 1 liter/day of one experimental beverage (containing 0.2% olive oil + 0.6% DHA-S Martek). Follow-up 8 weeks. At week 8 an acute exercise season was programed.
  One blood sample was taken in resting conditions at beginning of the nutritional intervention (week 0, baseline). Another two blood samples were taken at the end of the nutritional intervention, in resting (week 8, pre-exercise) and post-exercise conditions (week 8, post-exercise). Biochemical measures, oxidative damage markers on lipids, proteins and DNA, antioxidant capabilities (enzyme activities and quantity of enzyme protein and gene expression) and inflammatory markers were measured in serum, plasma, erythrocytes, neutrophils and peripheral blood mononuclear cells.
  Arms: Docosahexaenoic acid
Dietary Supplement: Placebo supplementation — Six professionals soccer players (19 and 22 years old) took 1 liter/day of placebo beverage (containing 0.8% olive oil). Follow-up 8 weeks. At week 8 an acute exercise season was programed.
  One blood sample was taken in resting conditions at beginning of the nutritional intervention (week 0, baseline). Another two blood samples were taken at the end of the nutritional intervention, in resting (week 8, pre-exercise) and post-exercise conditions (week 8, post-exercise). Biochemical measures, oxidative damage markers on lipids, proteins and DNA, antioxidant capabilities (enzyme activities and quantity of enzyme protein and gene expression) and inflammatory markers were measured in serum, plasma, erythrocytes, neutrophils and peripheral blood mononuclear cells.
  Arms: Olive oil

SUMMARY:
There are conflicting evidences of the effects of dietary supplementation with polyunsaturated fatty acids (PUFAs) on athletic performance. The investigators working hypothesis is based on the polyunsaturated fatty acids, given its pro-oxidative character and also by its action on transcription factors can modulate the antioxidant response and oxidative damage induced by physical activity.The overall objective of the study is to establish situations improving athletic performance and study the oxidative balance by manipulation of feeding patterns and consumption of nutritional supplements and investigate the involved mechanisms.

DETAILED DESCRIPTION:
There are conflicting evidences of the effects of dietary supplementation with polyunsaturated fatty acids (PUFAs) on athletic performance. The described effects of PUFAs on the fat metabolism may be modulated by the expression and activity of transcription factor genes, suppressing or expressing genes associated with the synthesis and oxidation of fats and in oxidative stress and inflammation.

The investigators' working hypothesis is based on the polyunsaturated fatty acids, given its pro-oxidative character and also by its action on transcription factors can modulate the antioxidant response and oxidative damage induced by physical activity.

In the field of professional sports and leisure use of food and / or antioxidants in the belief that these elements prevent muscle damage is very established. Most studies in athletes supplemented with antioxidant nutrients revealed no significant effects on physical performance, but it has shown that supplements protect against tissue damage induced by exercise. Recent studies have reported that over 35% of the Spanish people eat diets low or very low quality, which is clearly shown that over 10% of Spaniards have poor intakes (<2/3 IDR) riboflavin (men) , folate (women), vitamin C, vitamin A, vitamin D and vitamin E.

The overall objective of the study is to establish situations improving athletic performance and study the oxidative balance by manipulation of feeding patterns and consumption of nutritional supplements and investigate the involved mechanisms. The aim of this study is to establish scientific basis for design functional foods improving athletic performance and health and avoiding the negative consequences of the oxidative damage induced by overexertion.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 16 to 35 years
* Genders eligible for study: Male
* Equilibrate diet
* Physical activity of 1-2 hours daily 5-7 days weekly.
* Body mass index (19-25 kg/m2)

Exclusion Criteria:

* Smokers

Ages: 16 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
DHA incorporation in erythrocyte cellular membranes | Baseline, week 8
  Docosahexaenoic acid (DHA) is a conditionally essential fatty acid. Primary outcome: DHA incorporation in the erythrocyte cellular membranes by gas chromatography of soccer players during a training season

SECONDARY OUTCOMES:
DHA on oxidative stress | Baseline, week-8 (pre- and post-exercise)
  Effects of DHA diet supplementation, the training season and acute exercise on oxidative and nitrosative damage markers and antioxidant enzyme activities, and protein levels in different blood fractions.
DHA on inflammation | Baseline, week-8 (pre- and post-exercise)
  Effects of DHA diet supplementation, the training season and acute exercise on inflammation markers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Result] Capo X, Martorell M, Sureda A, Llompart I, Tur JA, Pons A. Diet supplementation with DHA-enriched food in football players during training season enhances the mitochondrial antioxidant capabilities in blood mononuclear cells. Eur J Nutr. 2015 Feb;54(1):35-49. doi: 10.1007/s00394-014-0683-2. Epub 2014 Mar 19. PMID 24643755
- [Result] Martorell M, Capo X, Sureda A, Tur JA, Pons A. Effects of docosahexaenoic acid diet supplementation, training, and acute exercise on oxidative balance in neutrophils. Appl Physiol Nutr Metab. 2014 Apr;39(4):446-57. doi: 10.1139/apnm-2013-0331. Epub 2013 Nov 4. PMID 24669986
- [Derived] Capo X, Martorell M, Sureda A, Tur JA, Pons A. Effects of dietary Docosahexaenoic, training and acute exercise on lipid mediators. J Int Soc Sports Nutr. 2016 Apr 5;13:16. doi: 10.1186/s12970-016-0126-y. eCollection 2016. PMID 27051354